CLINICAL TRIAL: NCT00592488
Title: Prospective, Randomized, Placebo-controlled, Double-Blinded, Phase II Pilot Study of Acetyl-L-carnitine in the Treatment of Patients With Septic Shock
Brief Title: Acetyl-L-Carnitine in the Treatment of Septic Shock
Acronym: ALC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Todd Rice, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 050730
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Results first posted 2011-06-08 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Septic Shock
Keywords: Septic shock; Acetyl-L-carnitine
MeSH Terms: conditions — Shock, Septic | interventions — Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Placebo for first 6 hours then Acetyl-L-Carnitine (ALC) for 12 hours
  Interventions: Drug: Acetyl-L-Carnitine
- B (Other): Acetyl-L-Carnitine (ALC) for first 12 hours then placebo for next 6 hours
  Interventions: Drug: Acetyl-L-Carnitine

INTERVENTIONS:
Drug: Acetyl-L-Carnitine — Acetyl-L-Carnitine - 4 g IV over 30 minutes, then 8 g iv over the next 12 hours
  Other Names: ALC

SUMMARY:
This placebo-controlled study investigates acetyl-L-carnitine in the treatment of septic shock requiring vasopressors.

DETAILED DESCRIPTION:
This is a cross-over study which infuses ALC for 12 out of 18 hours (and placebo the other 6). Patients must have vasopressor-dependent septic shock and be free from renal failure, hepatic failure, and seizures to be eligible.

ELIGIBILITY:
Inclusion Criteria:

* documented or presumed infection
* shock requiring vasopressors

Exclusion Criteria:

* dialysis
* hepatic failure
* seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-08; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd W. Rice, MD, MSc, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then ALC: Placebo for first 6 hours then ALC for 12 hours
- ALC Then Placebo: ALC for first 12 hours then placebo for next 6 hours
Period: Overall Study
Arm/Group | Placebo Then ALC | ALC Then Placebo
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then ALC | ALC Then Placebo | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Blood Pressure
Description: Mean Arterial blood pressure measured non-invasively at 18 hours
Time Frame: 18 hours
Population: All patients treated. Intention to treat.
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Acetyl-L-Carnitine (ALC) Then Placebo: ALC for hours 0-12 and placebo hours 12-18
- Placebo Then Acetyl-L-Carnitine (ALC): Placebo for hours 0-6 then ALC for hours 6-18
Arm/Group | Acetyl-L-Carnitine (ALC) Then Placebo | Placebo Then Acetyl-L-Carnitine (ALC)
Number analyzed (Participants) | 7 | 6
mm Hg | 60 (3) | 60 (4)

2. Secondary Outcome: Vasopressor Dose
Description: Change in vasopressor dose between 6 and 24 hours.
Time Frame: 6-24 hours
Measure: Mean (Standard Deviation); unit: mcg/kg/min
Groups:
- Placebo Then ALC: Placebo for first 6 hours then Acetyl-L-Carnitine (ALC) for 12 hours
  Acetyl-L-Carnitine: Acetyl-L-Carnitine - 4 g IV over 30 minutes, then 8 g iv over the next 12 hours
- ALC Then Placebo: Acetyl-L-Carnitine (ALC) for first 12 hours then placebo for next 6 hours
  Acetyl-L-Carnitine: Acetyl-L-Carnitine - 4 g IV over 30 minutes, then 8 g iv over the next 12 hours
Arm/Group | Placebo Then ALC | ALC Then Placebo
Number analyzed (Participants) | 7 | 6
mcg/kg/min | -1.4 (4.4) | -4.8 (5.9)

3. Secondary Outcome: Serum Lactate
Description: Latest serum lactate between 12 and 36 hours
Time Frame: 12-36 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Then ALC | ALC Then Placebo
Number analyzed (Participants) | 7 | 6
mg/dL | 2.1 (1.7) | 2.0 (1.8)

ADVERSE EVENTS:
Arm/Group | Placebo Then ALC | ALC Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No